CLINICAL TRIAL: NCT01278056
Title: The Impact of Deferasirox on Non-Alcoholic-Steatohepatitis (NASH) - a Prospective Open Label Phase I/II Trial
Brief Title: The Impact of Deferasirox on Non-Alcoholic-Steatohepatitis
Acronym: DEFINE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Crolll Gmbh (Other)
Collaborators: Estimate, GmbH (Industry); University of Magdeburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670EDE08T
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Non-alcoholic Steatohepatitis; Increased Iron Storage / Disturbed Distribution
Keywords: Non-alcoholic steatohepatitis (NASH) and increased iron storage / disturbed distribution
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exjade (Experimental)
  Interventions: Drug: Exjade

INTERVENTIONS:
Drug: Exjade — Two dose escalating cohorts of oral administration in Phase I. Phase II: oral administration of the maximum tolerated dose.
  Other Names: Deferasirox, ICL670

SUMMARY:
This is a Phase I/II open-label uncontrolled, prospective study to assess the clinical and biological effects of Deferasirox (ICL 670, Exjade®) in patients with NASH and increased iron storage / distribution of iron on liver function and liver histology.

NASH is defined clinically and histologically by elevated liver enzymes, signs of hepatic steatosis on ultrasound and magnetic resonance imaging, impaired liver function as expressed by functional breath tests, and significantly altered liver histology.

Patients will be treated in a phase I and phase II part for either 12 or 48 weeks.

Both study parts have different endpoints: in phase I the side effect profile will be evaluated while in phase II the therapeutic response will be tested. Accordingly, measures will be different.

Approximately 10 patients in phase I and 50 patients in phase II will be enrolled according to sample size calculations.

The design is an "adaptive" Two-stage design, allowing to minimize the number of patients included into the trial as well as to introduce corrections for the second stage.

ELIGIBILITY:
Inclusion Criteria (shortened):

* Patients with elevated liver enzymes
* Elevated serum ferritin (females > 300 ng/ml, males > 450 ng/ml)
* Liver Histology consistent with a diagnosis of NASH

Exclusion Criteria (shortened):

* Alcohol intake > 140 g/week
* Established liver cirrhosis Child Pugh B or C
* Copresence of other causes of chronic liver disease
* Anemia < 10 g/dl
* Any elevation of liver enzymes > 5 ULN (ALAT, ASAT, g-GT), > 2.5 ULN (other), > 1.5 (Bilirubin)
* Serum creatinine > 1.4 mg/dl or Ccr < 60 ml/min
* Hemochromatosis
* Known allergy or contraindication to the administration of Deferasirox
* Sexually active pre-menopausal female patients who are unable to use a highly effective method of birth control. An exception is made for those who have undergone clinically documented total hysterectomy and/or oophorectomy, tubal ligation.
* Patients with impaired coagulation
* History of blood transfusion during the 6 months prior to study entry
* Oral iron supplementation within the last 4 weeks of study entry
* Treatment with phlebotomy within 2 weeks of screening visit
* Desferal treatment within 1 month of the screening visit
* Patients currently or previously treated with deferiprone or Deferasirox
* Presence of a surgical or medical condition that might significantly alter the absorption, distribution, metabolism or excretion of any study drug
* Positive HIV serology
* Patients with active inflammatory diseases that may interfere with the accurate measurement of serum ferritin
* Patients with a diagnosis of a clinically relevant cataract or a previous history of clinically relevant ocular toxicity related to iron chelation
* Pregnant or breast feeding patients
* Patients treated with systemic investigational drug within 4 weeks prior or with topical investigational drug within 7 days prior to the screening visit
* Medications with proven or suspected influence on NASH such as glitazones, statins, or metformin are no exclusion criteria for study entry (insulin is not regarded to interfere with NASH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of deferasirox in all patients (Phase I) | Phase I: 12 weeks of treatment
  Safety and tolerability assessments will consist of evaluating (serious) adverse events, laboratory parameters including hematology, chemistry; vital signs and physical examinations according to CTC.
Changes in liver histology in all patients (Phase II) | Phase II: 48 weeks of treatment
  A decrease in the NASH activity score (NAS) of ≥1 compared to baseline will be classified as response, an unchanged score or an increase in NAS will be judged as non-response.

SECONDARY OUTCOMES:
Phase I: e.g. changes in liver enzymes, serum ferritin, and hemoglobin levels | Phase I: 12 weeks of treatment
Phase II: e.g. changes in MRI and histology based assessment of hepatic steatosis, fibrosis and iron content | Phase II: 48 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Treiber, PD Dr. med., Principal Investigator
Locations (9):
- Germany (9):
  - Zollernalbklinikum, Balingen/Hechingen
  - Charité, Virchow Klinikum, Berlin
  - Klinikum der J. W. Goethe-Universität, Med. Klinik I, Frankfurt
  - Universitätsklinikum Halle, Klinik & Poliklinik für Innere Medizin I, Halle
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Universitätsklinikum Magdeburg, Klinik für Gastroenterologie, Hepatologie und Infektiologie, Magdeburg
  - Universitätsklinikum Mainz, I. Medizinische Klinik und Poliklinik, Mainz
  - Universitätsklinikum Regensburg, Klinik und Poliklinik für Innere Med. I, Regensburg
  - Universitätsklinikum Tübingen, Medizinische Klinik IV, Tübingen